CLINICAL TRIAL: NCT06502470
Title: Open Label Study to Explore Healing and Tissue Histopathology Following Ellacor Micro-Coring Procedures in an Abdominoplasty Model
Brief Title: Healing Study of Fractional Skin Resurfacing and Tissue Histopathology After Ellacor Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cytrellis Biosystems, Inc. (Industry)
Collaborators: Dallas Plastic Surgery Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TP-00437
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Wrinkle; Rhytides; Histopathology
Keywords: Mechanism of Healing; Micro-Coring; Abdominoplasty; Histopathology; Immunohistochemistry; Wrinkle treatment; Fractional Skin Resurfacing

STUDY DESIGN:
Intervention Model Description: Abdominoplasty model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Safety Evaluation of Skin Removal Percentages and Evaluation of Healing over 14 Days. (Experimental): Three participants will have the ellacor® procedure done at 4 different timepoints before their abdominoplasty surgery: -14 days, -7 days, -3 days and on day 0, just prior to the abdominoplasty procedure. At each treatment timepoint the participants will have 3 areas treated using different skin removal percent settings: 5%, 7% and 8%. The participants will have photos taken of the treatment areas and will be asked about any changes to their health or medications over the 14-day study.
  Interventions: Device: ellacor® Micro-Coring procedure

INTERVENTIONS:
Device: ellacor® Micro-Coring procedure — ellacor® Micro-Coring Technology is FDA approved for use by medical professionals for the treatment of moderate and severe wrinkles in the mid and lower face in adults aged 22 years or older with Fitzpatrick skin types I-IV.

SUMMARY:
The goal of this study is to observe the healing of skin after ellacor® treatment at different timepoints, depths and coring densities. The visual comparison of treated areas to untreated control areas will improve understanding of how the ellacor® procedure works to induce skin resurfacing using an abdominoplasty, or tummy tuck surgery, model. The people participating in the study will have already decided that they want to have an abdominoplasty procedure.

The main questions this study aims to answer are:

How does human skin change after a series of the ellacor® procedures over a 14-day period?

Is the ellacor® device safe to use at different treatment time points, depths and densities?

The ellacor® procedure will be performed on people who are going to have abdominoplasty surgery. The ellacor® treatment areas will be limited to the skin areas marked for removal during the abdominoplasty. The treated tissue will be sent to a lab for microscopic study after the abdominoplasty procedure is complete. A minimum of 3 people will be treated in the study.

The 3 participants will have the ellacor® procedure done at 4 different timepoints before their abdominoplasty surgery: -14 days, -7 days, -3 days and on day 0, just prior to the abdominoplasty procedure. At each treatment timepoint the participants will have 3 areas treated using a depth of 7mm and different skin removal percent settings of 5%, 7% and 8%. The participants will have photos taken of the treatment areas and will be asked about any changes to their health or medications over the 14-day study.

Researchers will study the abdominoplasty tissue under a microscope after it has been removed from the participants. They will compare the areas treated by the ellacor® device to an area left untreated, which is the control area. This will reveal, by visual comparison, any changes in the skin tissue between treated and untreated areas, if they occur.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing planned abdominoplasty
* Are willing to donate their tissue for evaluation
* BMI ≤ 30
* Women 18 years or older
* Fitzpatrick scale I-VI
* Females of childbearing potential will have a negative urine pregnancy test prior to each procedure
* Are judged to be in good health based on the results of a medical history and physical examination (standard of care for abdominoplasty) at screening
* Has been informed of the nature of the study and agrees to its provisions and has provided written informed consent on a form, as approved by the IRB of the respective clinical site.
* Able and willing to comply with all visits, procedures and evaluation schedules and requirements

Exclusion Criteria:

* Having an active bleeding disorder or currently taking anticoagulants
* History of keloid formation or abnormal wound healing
* Inflammation or active infection and treatment area
* Compromised immune system (e.g., diabetes)
* Any surgery or treatments in the abdominal area 12 months prior to procedure
* Comorbid condition that could limit ability to participate in the study or to comply with follow up requirements
* Pregnant or breastfeeding
* Tattoo and/or mole located within the planned treatment area(s)
* Vulnerable populations include those defined 45 CFR 46 Subparts B, and those mentioned in 45 CFR 46.111(b): mentally disabled persons, or economically or educationally disadvantaged persons
* Any issue that at the discretion of the investigator would contraindicate the subject's participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 3 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Adverse events will be collected from Day 0 (the initial ellacor treatment day) through the day of the scheduled abdominoplasty procedure (Day 14 for all subjects).
  The incidence and severity of adverse events will be evaluated for all subjects enrolled to the study.
The change in histopathology of abdominoplasty tissue samples after sequential treatments with the ellacor® device at a micro-coring depth of 7mm over a 14-day period as compared to an untreated control area. | The abdominoplasty tissue will be excised 14 days after the initial ellacor® treatment. Histopathological studies will be performed upon receipt at the central pathology laboratory.
  This 14-day healing evaluation of fractional skin resurfacing will compare the histopathology of stained tissue isolated after sequential ellacor® treatments on abdominal skin tissue. The samples will be isolated from excised abdominal tissue following abdominoplasty. The tissue will include an untreated control area compared to three ellacor® treated areas with depth of treatment at 7mm and different tissue percentage removal settings. Area 1 = 5% tissue removal, Area 2 = 7% and Area 3 = 8%. Each area will be treated on Day -14, Day -7, Day -3 and Day 0, the day of abdominoplasty. Histopathological evaluation will include Hematoxylin and Eosin (H&E), Herovici, and Movat stains. The stains will provide comparison of structural tissue changes (H&E stain), change in presence of Type III (young) collagen and Type I (mature) collagen (Herovici stain) and change in presence of collagen, fibrin and elastic fibers (Movat stain) over the 14-day time period compared to untreated control area.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Edgecombe, Study Director — Cytrellis Biosystems, Inc.
Locations (1):
- Dallas Plastic Surgery Institute, Dallas, Texas, United States